CLINICAL TRIAL: NCT04220424
Title: Glioma Patients Registry Based on MR Images, Histopathology Images and Genetic Sequencing Analyzed by Artificial Intelligence
Brief Title: Glioma Patients Registry Based on Radiological, Histopathological and Genetic Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Principal Investigator, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: GliomaAI-6
Record Dates: First submitted 2020-01-04; First posted 2020-01-07 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Glioma
Keywords: Artificial intelligence; MR images; histopathology images; sequencing; mechanism
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — All participants have signed the informed consent. Fresh frozen tissues of participants are collected immediately after tumor resection and preserved in liquid nitrogen. Whole exome sequencing, RNA sequencing and proteomics,etc are planed to be conducted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MR and Histopathology images based prediction of molecular pathology and patient survival — MR and Histopathology images based prediction of molecular pathology and patient survival in gliomas by leverage artificial intelligence algorithms

SUMMARY:
This prospective study aims to collect clinical, radiological, pathological, molecular and genetic data including detailed clinical parameters, MR and histopathology images, molecular pathology and genetic sequencing data. By leveraging artificial intelligence, this registry seeks to construct and refine algorithms that able to predict molecular pathology or clinical outcomes of glioma patients based on MR images and histopathology images, as well as revealing related mechanisms from genetic perspective.

DETAILED DESCRIPTION:
Non-invasive and precise prediction for molecular biomarkers such as 1p/19q co-deletion, MGMT methylation, IDH and TERTp mutations, and patients survival is challenging for gliomas. With the development of artificial intelligence, much more potential lies in the preoperative conventional/advanced MR imaging (T1 weighted imaging, T2 weighted imaging, FLAIR, contrast-enhanced T1 weighted imaging, diffusion-weighted imaging, and perfusion imaging), and in the histopathology images of HE slices of gliomas could be excavated to aid prediction of molecular pathology and patients' survival of gliomas. This study aims to collect clinical, radiological, pathological, molecular and genetic data including detailed clinical parameters, MR and histopathology images, molecular pathology (1p/19q co-deletion, MGMT methylation, IDH and TERTp mutations, etc) and genetic data (Whole exome sequencing, RNA sequencing, proteomics, etc), and seeks to construct and refine algorithms that able to predict molecular pathology or clinical outcomes of glioma patients based on MR images and histopathology images, as well as revealing related mechanisms from genetic perspective.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiologically and histologically confirmed diagnosis of primary glioma
* Life expectancy of greater than 3 months
* Must receive tumor resection
* Must have sufficient frozen tissues and peripheral blood samples for sequencing
* Must have high-quality MR images and histopathology images
* Signed informed consent

Exclusion Criteria:

* No gliomas
* No sufficient amount of tumor tissues for detection of molecular pathology
* Patients who are pregnant or breast feeding
* Patients who are suffered from severe systematic malfunctions

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed glioma that receive tumor resection with preoperative MR images and postoperative histopathology images
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
AUC of Prediction performance | up to 2 years
  AUC of Prediction performance=sensitivity+specificity-1

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided